CLINICAL TRIAL: NCT05646433
Title: Validation of a New Tunisian Risk Score for Upper Gastrointestinal Bleeding in the Emergency Room: Study of the TU-GIB Score
Brief Title: Validation of a New Score for UGI Bleeding in the ED: the Study of the TU-GIB Score
Acronym: TU-GIBscore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, clinical professor, Hôpital Universitaire Sahloul
Other Study IDs: TU-GIBscore
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Gastro Intestinal Bleed
Keywords: Upper Gastro intestinal bleeding; TU-GIB score; ED
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We have developed a new reliable, easy and reproducible clinical and biological score to select patients presenting to the emergency department with upper GI bleeding and at high risk of developing complications in order to plan an adequate management.

This score was compared to the Glasgow-Blatchford score and showed better results in predicting rebleeding, the need for hemostasis therapy and any complications at day 30 including mortality.

In a second step and as an objective of this study, it is necessary to perform an external validation of this score in different emergency departments.

DETAILED DESCRIPTION:
We have developed a new reliable, easy and reproducible clinical and biological score to select patients presenting to the emergency department with upper GI bleeding and at high risk of developing complications in order to plan an adequate management.

This score was compared to the Glasgow-Blatchford score and showed better results in predicting rebleeding, the need for hemostasis therapy and any complications at day 30 including mortality.

In a second step and as an objective of this study, it is necessary to perform an external validation of this score in different emergency departments.

We will conduct a multicenter, descriptive and analytical study in different emergency departments Inclusion criteria: patients consulting the emergency department for upper GI hemorrhage of non-traumatic origin.

Exclusion criteria: patients under 18 years of age, diagnosed with external hemorrhoids with parietal lesions. We exclude any patient who does not consent, is lost to follow-up or has incomplete information.

Anonymity and confidentiality of the data were respected. Data collection was carried out using a data processing form designed for the purpose of this work, including descriptive analysis of the epidemiological and clinical characteristics of the patients, as well as the para-clinical data.

Patients were followed up by telephone call at D30 to record the date and cause of any complications noted, such as rebleeding, hospitalization, or death.

The data will be entered and analyzed in SPSS 21.0

ELIGIBILITY:
Inclusion Criteria:

* patients consulting the emergency room for upper GI hemorrhage of non-traumatic origin.
* Age >18 years

Exclusion Criteria:

* patient under the age of 18
* Lower gastrointestinal hemorrhag
* diagnosis of external hemorrhoids / perianal lesions
* Not consenting
* The lost sight

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multicentric, descriptive and analytical study in different emergency departments
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was all-cause in-hospital mortality rate | 30 days after inclusion
  The primary outcome was all-cause in-hospital mortality rate

SECONDARY OUTCOMES:
re-bleeding, re-hospitalization, discharge | 30 days after inclusion
  Hemorrhagic recurrence is defined by recurrence of hematemesis, melena or rectal bleeding after discharge from hospital within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sahloul University Hospital, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided